CLINICAL TRIAL: NCT07267949
Title: Clinical Randomised Phase 2 Trial of AP31969 Versus Placebo for Rhythm Control of Atrial Fibrillation
Acronym: END-AF-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Acesion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP31969-M201; 2025-521377-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; AP31969; SK channel inhibitor
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Also the blinded CRO team will not be made aware of the treatment group assignment during the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AP31969 100 mg (Experimental): Tablets, Twice daily, 12 Weeks
  Interventions: Drug: AP31969
- AP31969 200 mg (Experimental): Tablets, Twice daily, 12 Weeks
  Interventions: Drug: AP31969
- AP31969 350 mg (Experimental): Tablets, Twice daily, 12 Weeks
  Interventions: Drug: AP31969
- AP31969 500 mg (Experimental): Tablets, Twice daily, 12 Weeks
  Interventions: Drug: AP31969
- Placebo (Placebo Comparator): Tablets, Twice daily, 12 Weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP31969 — Tablets, Oral, Twice daily.
  Arms: AP31969 100 mg; AP31969 200 mg; AP31969 350 mg; AP31969 500 mg
Drug: Placebo — Tablets, oral, Twice daily.
  Arms: Placebo

SUMMARY:
A clinical Randomized Phase 2 Trial of AP31969 versus Placebo for Rhythm Control of Atrial Fibrillation.

DETAILED DESCRIPTION:
The key goal of this clinical trial is to assess the effectiveness of different doses of AP31969 in lowering Atrial Fibrillation (AF) burden and its safety.

Participants will be randomly assigned to one of the following groups:

* AP31969 at 100 mg, 200 mg, or 350 mg doses
* AP31969 500 mg (not included at the trial start)
* Placebo (inactive treatment and has no active properties). The placebo group serves as the comparator for AP31969. All treatments are given orally, twice daily.

The trial includes 3 periods: screening (up to 4 weeks), treatment (12 weeks), and follow-up (30 days). The duration of the trial for a participant is approximately 20 weeks.

Participants will receive an implantable loop recorder and undergo assessments during the visits at specific times, for example blood and urine analyses, and electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Age 18 or older.
* ECG documented diagnosis of paroxysmal or persistent AF.
* AF history at screening indicating an expected AF burden of 1-90%, i.e., at least 1 self-terminating AF episode within 4 months prior to the screening visit.
* AF burden of ≥ 1% and ≤ 90% assessed with an ECG patch device during the screening period prior to the randomisation visit.
* Investigator and participant agreement to avoid non-trial related rhythm control intervention for the duration of the trial, including:

  * Antiarrhythmic drug class I and/or III (including amiodarone)
  * Electrical or pharmacological cardioversion
  * AF ablation procedure
* Willing to have a loop recorder implanted.

Exclusion Criteria:

* Prior AF ablation procedure other than pulmonary vein isolation (PVI) only.
* Any of the following events within 4 weeks prior to the screening visit: Myocardial infarction, Unstable angina pectoris, Stroke or transient, ischaemic attack, Percutaneous coronary intervention (PCI), Coronary artery bypass graft (CABG), Peripheral revascularisation procedure.
* Cardiac pacing device e.g. pacemaker and cardiac resynchronization therapy device with atrial or ventricular pacing for > 5% of the time or existing implantable loop recorder.
* Heart failure, New York Heart Association class III (3) or IV (4).
* Left ventricular ejection fraction < 40% based on imaging (e.g. echocardiography) performed within 6 months prior to or during the screening visit.
* Clinically significant valvular heart disease, including severe aortic stenosis, severe mitral regurgitation and/or severe mitral stenosis, in the opinion of the investigator.
* QTc (Fridericia, QTcF) interval > 450 ms for males and > 470 ms for females at screening.
* eGFR <60 mL/min /1.73 m² based on creatine and CKD-EPI formula
* Use of antiarrhythmic drug class I and/or III within 7 days or, for amiodarone, within 3 months prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden | From week 2 to week 12
  Measured through implantable loop recorder. Calculated as the amount of time with AF relative to the amount of time the participant is under observation (expressed as a %).

SECONDARY OUTCOMES:
Number of atrial fibrillation episodes | From week 2 to week 12
  Measured through implantable loop recorder.
Change from baseline in Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) | Week 12
  Patient reported outcome.
Number of ventricular tachycardia episodes > 30 seconds of duration | From week 0 to week 12
  Measured through implantable loop recorder.

CONTACTS AND LOCATIONS:
Locations (38):
- Bulgaria (6):
  - UMHAT "Sveti Georgi" EAD, Department of Invasive Cardiology, Plovdiv, PD
  - Acibadem City Clinic, Cardiology Department, Sofia, SOF
  - MHAT National Cardiology Hospital EAD, Cardiology Department, Sofia, SOF
  - Aleksandrovska University Hospital, Clinic of Cardiology, Sofia, SOF
  - SHATC Cardiolife, Invasive Cardiology, Varna, VAR
  - Medical Center Nova Clinic, Varna, VAR
- Denmark (2):
  - University Hospital Herlev and Gentofte Department of Cardiology, Hellerup
  - Viborg Hospital, Department of Cardiology, Viborg
- Germany (3):
  - Sana Kliniken Oberfranken, Klinikum Coburg Kardiologie und Innere Medizin, Coburg
  - Universitätsklinikum Frankfurt Medizinische Klinik III - Kardiologie, Angiologie, Hämostaseologie, Nephrologie, Frankfurt
  - Universitaets Klinikum Hamburg-Eppendorf (UKE Hamburg), Kardiologie, Hamburg
- Hungary (6):
  - Budai Irgalmasrendi Kórház, Budapest
  - Semmelweis Egyetem Városmajori Sziv- és Érsebészeti Klinika, Budapest
  - Soproni Gyógyközpont Soproni Erzsébet Oktató Kórház és Rehabilitációs Intézet, Sopron
  - Szent-Györgyi Albert Klinikai Központ, Belgyógyászati Klinika, Szeged
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház-Rendelőintézet, Szolnok
  - Belvárosi Egészségház, Platán Magánklinika, Zalaegerszeg
- Italy (5):
  - Policlinico Sant'Orsola Cardiology Department, Bologna, BO
  - Arcispedale Sant'Anna, Cardiology Department, Cona, FE
  - ASST Grande Ospedale Metropolitano Niguarda Cardiology 3 - Electrophysiology "De Gasperis" Cardio Center, Milan, Michigan
  - University of Modena and Reggio Emilia, Policlinico di Modena, Cardiology Department, Modena, Missouri
  - Dell'Angelo Hospital, Cardiology Department, Mestre, VE
- Netherlands (9):
  - Rijnstate Ziekenhuis, Cardiology Department, Arnhem
  - Deventer Ziekenhuis, Cardiology Department, Deventer
  - Martini Hospital Groningen, Cardiology Department, Groningen
  - Spaarne Gasthuis, Cardiology Department, Haarlem
  - Frisius MC Leeuwarden, Hart- en Vaatcentrum, Leeuwarden
  - Maastricht University Medical Center, Cardiology Department, Maastricht
  - HagaZiekenhuis, Cardiology/Electrophysiology Unit, The Hague
  - Rivierenland Hospital, Cardiology Department, Tiel
  - Máxima Medisch Centrum, Cardiology Department, Veldhoven
- Poland (7):
  - Centrum Medyczne KERmed Cardiology Department, Bydgoszcz
  - Małopolskie Centrum Sercowo-Naczyniowe PAKS Oddział Intensywnej Opieki Kardiologicznej, Chrzanów
  - Polsko-Amerykańskie Kliniki Serca III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii, Dąbrowa Górnicza
  - Gornoslaskie Centrum Medyczne im. prof. Leszka Gieca Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Upper-Silesian Medical Center 2nd Department of Cardiology, Katowice
  - One Day Med Sp. z o.o. Clinical Trials Department, Szczecin
  - Polsko-Amerykańskie Kliniki Serca X Oddział Kardiologii Inwazyjnej, Elektrofizjologii i Elektrostymulacji w Tychach im, Tychy

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request access to anonymized data and needed trial documentation. Requests are evaluated on the basis of scientific merit. Any use of and access to the data must respect the privacy of the participants and will only be provided if applicable laws and regulations allow this.